CLINICAL TRIAL: NCT01304628
Title: A Phase 2a, Double-Blinded, Multi-Center, Escalating Dose Group, Placebo Controlled, Cross-Over Study to Evaluate the Safety, Efficacy and Tolerability of Subcutaneously Administered PL-3994 for the Treatment of Patients With Mild to Moderate Asthma
Brief Title: Cross-Over Study of Subcutaneous Study Drug for the Treatment of Patients With Mild to Moderate Asthma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study prior to initiation.
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PL-3994-501
Record Dates: First submitted 2011-02-22; First posted 2011-02-25 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — PL-3994

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PL-3994 (4 escalating doses) (Experimental)
  Interventions: Drug: PL-3994
- Placebo (Placebo Comparator)
  Interventions: Drug: PL-3994

INTERVENTIONS:
Drug: PL-3994 — subcutaneous PL-3994, single dose, 4 escalating dose groups

SUMMARY:
The objective of this study is to evaluate if single subcutaneous (SC) doses of PL-3994, administered to patients with asthma can achieve a clinically meaningful increase in pulmonary function (Forced Expiratory Volume in one second: FEV1) while maintaining an acceptable safety profile. The study will characterize the bronchodilator effect, dose and safety of PL-3994 in a population of moderately severe, stable asthmatics following overnight withdrawal of beta-2 agonists.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent
* The subject is male or female >18 to 65 years of age
* Patient has a clinical history of asthma as defined by the National Asthma Education and Prevention Program.
* Documented bronchodilator response to albuterol as defined by the American Thoracic Society (> 200 mL and > 12% increase in FEV1 after bronchodilator inhalation)
* FEV1 post-bronchodilator of between 55% and 80% predicted.
* Currently taking 200-1000 mcg (fluticasone equivalent) of inhaled corticosteroids
* All inclusion criteria met within the past 12 months.
* If the subject or subject's partner is of child-bearing potential, a medically acceptable form of contraception will be used for three months prior to the screening visit (females only), for the duration of the study and for one month following the last dose of the study drug. Medically acceptable contraceptives include: (1) surgical sterilization, (2) FDA-approved female hormonal contraceptives, (3) an intrauterine device (IUD), (4) condoms with spermicide, or (5) diaphragm with spermicide.

If the subject had a vasectomy greater than 6 months prior to the screen visit, this will also be acceptable.

Exclusion Criteria:

* Current diagnosis, as per subject or investigator or screening assessment, of:

  * unstable or uncontrolled disease in any organ system (including cardiovascular) on present therapy
  * psychiatric disease requiring daily medication, including controlled or uncontrolled schizophrenia or any other uncontrolled psychiatric condition
  * significant neurological disease
  * current or history of any cancer (except non-melanomatous skin cancer) diagnosed less than 5 years prior to screening
  * acute or chronic disease requiring frequent changes in medications or changes in dosages of chronic therapy
  * history of alcohol abuse within the past 5 years
  * positive result for the alcohol and/or drug tests at screening or check-in
  * positive for HIV, or Hep B&C at screening
  * blood donation within 30 days of screening or plasma donation within 7 days of screening
  * weight > 100 kg or < 50 kg
  * clinically significant electrocardiogram (ECG) at screening
  * any clinically significant (per the investigator) lab abnormalities
  * any fever or other clinically significant physical exam abnormalities
* History of COPD or any other lung disease
* Greater than 10 packs per year smoking history and any cigarette smoking within the past 12 months
* Patients unable to withhold bronchodilator treatment for 12 hours prior to dosing
* Patients with hypoxia at screen or Check -in Visit 2, Day 1 or Visit 3, Day 7 (oxygen saturation measured by pulse oximetry [SpO2] < 90%)
* Tachycardia (heart rate > 100 beats/min) at screening
* Currently being treated for Hypertension or taking any other medications that affect blood pressure significantly.
* Currently taking any medications that inhibit PDE activity or which affect the cyclic guanisine mono-phosphate (cGMP) pathway (e.g. theophylline). These medications will be prohibited during the study and for at least 5 half- lives prior to Check-in Visit 2, Day 1 or Visit 3, Day 7 so that cGMP measurements will not be affected.
* Hypotension (systolic blood pressure < 110 mmHg) at Screening or Check-in Visit 2, Day 1 or Visit 3, Day 7
* Chronic kidney disease defined as estimated glomerular filtration rate (eGFR) <50 mL/m2.
* Diagnosis of heart failure or history of hospitalization for congestive heart failure.
* History of coronary artery disease defined as prior myocardial infarction, prior revascularization procedure, or >50% coronary artery obstruction by angiography.
* Prior history of stroke or transient ischemic attack.
* Female patients of childbearing potential who are nursing or have a positive pregnancy test at Screening or Check -in Visit 2, Day 1 or Visit 3, Day 7
* Any major disability or disease with expected survival less than 6 months
* Administration of any investigational drug or implantation of investigational device, or participation in another trial, within 30 days of screening.
* Inability to perform acceptable, quality serial spirometry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in one second (FEV1) | Throughout 12 hours post dosing
  Serial spirometry measures, including FEV1, assessed at specified time periods over 12 hours post dose.

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Throughout 12 hours post dosing
  Serial spirometry measures, including FVC, assessed at specified time periods over 12 hours post dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Cranbury, New Jersey, United States